CLINICAL TRIAL: NCT00230074
Title: A Long-term Extension Study of TCH346 and Placebo Administered Once Daily in Patients With Amyotrophic Lateral Sclerosis(ALS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTCH346A2211E1
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — dibenzo(b,f)oxepin-10-ylmethyl-methyl-prop-2-ynyl-amine

INTERVENTIONS:
Drug: TCH346

SUMMARY:
This is a study to evaluate the safety and clinical effects of 4 oral doses of TCH346 compared to placebo in patients with mild or mild to moderate stages of ALS.

DETAILED DESCRIPTION:
This is a study to evaluate the safety and clinical effects of 4 oral doses of TCH346 compared to placebo in patients with mild or mild to moderate stages of ALS.

ELIGIBILITY:
Inclusion Criteria:

* Completed original protocol, Study No. CTCH346A2211
* Be capable of satisfying the requirements of the extension protocol and must sign informed consent after the nature of the extension protocol has been fully explained

Exclusion Criteria:

* Exclusion criteria as described in the original protocol will remain applicable into the extension protocol

Other protocol-defined exclusion criteria may apply.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2004-11; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Rate of functional decline as defined by the ALS Functional Rating Scale-Revised

SECONDARY OUTCOMES:
Survival time
Functional outcome measures including pulmonary function and manual muscle strength assessments (every visit)

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis, East Hanover, New Jersey, United States